CLINICAL TRIAL: NCT03163472
Title: A Comparison of the Effects of Two Volumes (10 vs 30 mL) of Lidocaine 2% With Epinephrine 1:200 000 on the Duration of Ultrasound Guided Axillary Brachial Plexus Block.
Brief Title: Effect of Local Anaesthetic Volume on Axillary Brachial Plexus Block Duration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cork University Hospital (Other)
Responsible Party: Principal Investigator, Dr Anil Ranganath, Dr (Fellow in Regional Anaesthesia), Cork University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ECM 4 (J)
Record Dates: First submitted 2017-05-07; First posted 2017-05-23 (Actual); Results first posted 2021-08-31 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Brachial Plexus Blockade
MeSH Terms: interventions — Anesthesia, Local

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10 ml of lidocaine 2% with epinephrine (Active Comparator): patients will receive axillary brachial plexus block with 10 ml of lidocaine 2% with epinephrine.
  Interventions: Procedure: Axillary brachial plexus block with 10 mL oof local anaesthetic
- 30ml of lidocaine 2% with epinephrine (Experimental): patients will receive axillary brachial plexus block with 30 ml of lidocaine 2% with epinephrine.
  Interventions: Procedure: Axillary brachial plexus block with 30 ml of local anaesthetic

INTERVENTIONS:
Procedure: Axillary brachial plexus block with 10 mL oof local anaesthetic — patients will receive axillary brachial plexus block with 10 ml of lidocaine 2% with epinephrine.
  Arms: 10 ml of lidocaine 2% with epinephrine
Procedure: Axillary brachial plexus block with 30 ml of local anaesthetic — patients will receive axillary brachial plexus block with 30 ml of lidocaine 2% with epinephrine.
  Arms: 30ml of lidocaine 2% with epinephrine

SUMMARY:
Axillary brachial plexus block is an safe, effective and widely used technique for providing surgical anesthesia at and below the elbow. Inadvertent intraneural and intravascular injections are the only significant risks. Traditionally, greater volumes of local anaesthetic have been administered to achieve successful axillary brachial plexus block, but recent studies have demonstrated that this can be achieved with even very low volumes of 2-4 mL lidocaine 1.5% per nerve or ultra low volume of 1 mL lidocaine 2% per nerve.

Administration of 30mL (vs 10 mL) lidocaine 2% with epinephrine 1:200 000 prolongs the sensory and motor block duration of ultrasound guided axillary brachial plexus block for elective upper limb surgical procedures.

Primary Outcome:

The primary outcome will be the overall duration of sensory block.

Secondary Outcomes:

Duration of motor block Time to onset of the block. The quality of block intraoperatively Time to first request of postoperative opioid analgesia. Total opioid consumption at 24 hours. The incidence of adverse effects perioperatively: nausea, dizziness, tinnitus, vomiting, convulsions or arrhythmia.

DETAILED DESCRIPTION:
Peripheral nerve blocks provide significant benefits to patients, including improved analgesia and decrease in general anaesthesia-related adverse effects. Ideally peripheral nerve block provides rapid onset and substantial perioperative analgesia. Use of ultrasound guidance in peripheral nerve blocks offers significant advantages compared to alternative techniques. It improves block success rate and shortens onset time.

To compare the effects of local anaesthetic volumes (10 vs 30 mL) of lidocaine 2% with epinephrine 1:200 000 on the duration of sensory and motor block following ultrasound guided axillary brachial plexus block.

Methods:

It is a prospective, randomized, observer blinded study. With institutional ethical approval and having obtained written informed consent from each, 30 patients will be studied.

Randomization and blinding:

Using a computer generated and sealed envelope technique, 30 patients will be randomly allocated in to one of two groups.

Group 1: patients will receive 10 ml of lidocaine 2% with epinephrine. Group 2: patients will receive 30 ml of lidocaine 2% with epinephrine.

Sample size and statistical analysis:

Sample size calculation will be based on duration of sensory block as the primary outcome parameter. Kaabachi et al found a sensory duration of axillary brachial plexus block (with 30 mL of lidocaine 1.5%) of 126 (SD=48) mins. The minimum sample size required to have a 90% probability of detecting a decrease in duration of 60 mins (level of significance 0.05) will be 13 patients per group using an unpaired student's t test. Total recruited 30.

Anaesthetic procedure:

Having established intravenous access, standard anaesthetic monitoring will be applied. Premedication with midazolam will be administered as clinically indicated (to a maximum of 3 mg). The operative arm will be abducted and externally rotated with elbow flexed at 90 degrees. Under strict aseptic condition, ultrasound guided axillary brachial plexus block will be performed. Having identified musculocutaneous, median, radial and ulnar nerves, a 50mm 22-gauge ultraplex short bevel insulated needle will be used with in-plane approach to block each nerve with either 2.5 ml (10 mL group) or 7.5 ml (30 mL group). All blocks will be performed by single operator experienced in the ultrasound peripheral nerve blocks.

Block assessment:

When the block procedure has been completed, a blinded observer will assess the onset of sensory and motor block15 in the innervation of each nerve every 5 mins, until surgical anesthesia is achieved or 30 mins have elapsed. Surgical anesthesia will be defined as a motor score ≤2, with absent sensation to cold and pinprick. Each nerve distribution will be individually assessed. Onset time will be measured from conclusion of the block (t=0) to attainment of surgical anesthesia. Block will be deemed failure if surgical anesthesia has not been achieved at 30 mins in one or more of the four nerve distribution. In case of failure, an additional rescue block or conversion to general anesthesia will be performed. Data from these patients will be analysed separately.

Intraoperative period:

All patients will receive 1 g of paracetamol and diclofenac 75 mg iv during surgery. In case of patients discomfort sedation and rescue analgesia in the form of fentanyl 25 micrograms aliquots IV will be administered to a maximum of 100 micrograms.

Postoperative period:

Upon arrival to recovery room, sensory and motor function will be assessed every 15 mins by a blinded observer.15 Assessment will be performed for each nerve separately. Block regression is defined as a return of sensation to cold and pinprick with motor power score ≥3 in any nerve region. Time to first request of postoperative analgesia and total opioid consumption for 24 hrs will be noted. Postoperative analgesia will be prescribed as paracetamol 1 g 6 hourly and diclofenac sodium 75 mg 12 hourly. Oxycodone 5-10 mg orally 4-6 hourly will be administered as rescue analgesia.

Primary Outcome:

The primary outcome will be the overall duration of sensory block.

Secondary Outcomes:

Duration of motor block Time to onset of the block. The quality of block intraoperatively Time to first request of postoperative opioid analgesia. Total opioid consumption at 24 hours. The incidence of adverse effects perioperatively: nausea, dizziness, tinnitus, vomiting, convulsions or arrhythmia.

ELIGIBILITY:
Inclusion Criteria

* ASA 1-3
* Patients aged >18 years
* undergoing elective upper limb (forearm, wrist or hand) surgical procedures.

Exclusion Criteria

* Contraindications to regional anaesthesia
* Hypersensitivity to amide local anaesthetics.
* Chronic pain
* Language barrier
* Neuromuscular disorders or peripheral neuropathy
* Body mass index > 35
* History of hepatic and renal insufficiency
* Pregnancy
* Cognitive or psychiatric disorder
* Cardiac conduction abnormality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-11-14 (Actual); Primary Completion 2013-08-07 (Actual); Study Completion 2013-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anil Ranganath, FCAI, Principal Investigator — Cork University Hospital

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Assessed for eligibility: n= 60
  Excluded : n=30
  * Not meeting inclusion criteria: n = 5
  * Declined to participate: n= 25
Groups:
- 10ml of Lidocaine 2% With Epinephrine: patients will receive axillary brachial plexus block with 10 ml of lidocaine 2% with epinephrine.
  Axillary brachial plexus block: patients will receive axillary brachial plexus block with 10 ml of lidocaine 2% with epinephrine.
- 30ml of Lidocaine 2% With Epinephrine: patients will receive axillary brachial plexus block with 30 ml of lidocaine 2% with epinephrine.
  Axillary brachial plexus block: patients will receive axillary brachial plexus block with 30 ml of lidocaine 2% with epinephrine.
Period: Overall Study
Arm/Group | 10ml of Lidocaine 2% With Epinephrine | 30ml of Lidocaine 2% With Epinephrine
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 10 ml of Lidocaine 2% With Epinephrine: patients will receive axillary brachial plexus block with 10 ml of lidocaine 2% with epinephrine.
  Axillary brachial plexus block: patients will receive axillary brachial plexus block with 10 ml of lidocaine 2% with epinephrine.
- Total: Total of all reporting groups
Arm/Group | 10 ml of Lidocaine 2% With Epinephrine | 30ml of Lidocaine 2% With Epinephrine | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (15.1) | 50 (22.1) | 49.3 (18.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Overall Duration of Sensory Block.
Description: Duration of sensory block of ultrasound guided brachial plexus block
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | 10 ml of Lidocaine 2% With Epinephrine | 30ml of Lidocaine 2% With Epinephrine
Number analyzed (Participants) | 15 | 15
minutes | 165 [142 to 172] | 188 [173 to 205]
Statistical Analysis 1: Comparison: 10 ml of Lidocaine 2% With Epinephrine vs 30ml of Lidocaine 2% With Epinephrine; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Duration of Motor Block
Description: The total duration of motor block
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | 10 ml of Lidocaine 2% With Epinephrine | 30ml of Lidocaine 2% With Epinephrine
Number analyzed (Participants) | 15 | 15
minutes | 165 [147 to 180] | 195 [175 to 220]
Statistical Analysis 1: Comparison: 10 ml of Lidocaine 2% With Epinephrine vs 30ml of Lidocaine 2% With Epinephrine; Test type: Other; p = 0.001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Time to Onset of the Block
Description: Time to overall onset time for block
Time Frame: 6 hours
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | 10ml of Lidocaine 2% With Epinephrine | 30ml of Lidocaine 2% With Epinephrine
Number analyzed (Participants) | 15 | 15
minutes | 15 [10 to 15] | 10 [5 to 15]
Statistical Analysis 1: Comparison: 10ml of Lidocaine 2% With Epinephrine vs 30ml of Lidocaine 2% With Epinephrine; Test type: Other; p = 0.022, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Time to First Request of Postoperative Opioid Analgesia
Description: Post-operative, Time to first request of opioid analgesia by the participants
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | 10ml of Lidocaine 2% With Epinephrine | 30ml of Lidocaine 2% With Epinephrine
Number analyzed (Participants) | 15 | 15
minutes | 188 [168 to 224] | 267 [224 to 313]
Statistical Analysis 1: Comparison: 10ml of Lidocaine 2% With Epinephrine vs 30ml of Lidocaine 2% With Epinephrine; Test type: Other; p = 0.011, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Opioid Consumption
Description: overall cumulative opioid consumption dose of the participants
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | 10ml of Lidocaine 2% With Epinephrine | 30ml of Lidocaine 2% With Epinephrine
Number analyzed (Participants) | 15 | 15
mg | 8.3 (5.6) | 6.3 (6.9)

6. Secondary Outcome: Number of Participants With Adverse Effects Perioperatively: Nausea, Dizziness, Tinnitus, Vomiting, Convulsions or Arrhythmia"
Description: We recorded the the number of participants with adverse effects like nausea, dizziness, tinnitus, vomiting, convulsions or arrhythmia during the perioperative period.
Time Frame: 24 hours
Population: No adverse events noted in any participants in either group
Measure: Count of Participants; unit: Participants
Arm/Group | 10 ml of Lidocaine 2% With Epinephrine | 30ml of Lidocaine 2% With Epinephrine
Number analyzed (Participants) | 15 | 15
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 hours
Description: The Incidence of Adverse Effects peri-operatively: Nausea, Dizziness, Tinnitus, Vomiting, Convulsions or Arrythmia
Arm/Group | 10ml of Lidocaine 2% With Epinephrine | 30ml of Lidocaine 2% With Epinephrine
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No